CLINICAL TRIAL: NCT01090856
Title: Predilation of Side Branch During Percutaneous Treatment of Bifurcation Lesions With Provisional T Stenting.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PI 0209/09
Record Dates: First submitted 2010-03-22; First posted 2010-03-23 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Angiography
Keywords: Bifurcations; Drug eluting-stents; Provisional stenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No pre-dilation side branch (No Intervention)
- Pre-dilation side branch (Active Comparator)
  Interventions: Procedure: Pre-dilation side branch

INTERVENTIONS:
Procedure: Pre-dilation side branch — Balloon pre-dilation of the side branch to facilitate the ulterior wire access.
  Arms: Pre-dilation side branch

SUMMARY:
Percutaneous treatment of bifurcation lesion is a complex procedure. After main vessel stent implantation, the side branch became jailed and the carina can be displaced resulting in complete occlusion of this vessel. Re-wiring the side branch in this conditions may result difficult and some times impossible. There is no agreement regarding the need of side branch pre-dilation (before main vessel stent implantation) to reduce these complications. Researchers from European Bifurcation Club have proposed no to pre-dilate the side branch to avoid vessel dissection and difficulties in rewiring the true lumen of the vessel. On the contrary, our group has a good experience in the treatment of bifurcation lesions treated with side branch pre-dilation.

Aims: 1.- To determine the efficacy of the side-branch pre-dilation in patients with bifurcations lesions treated with provisional T stenting. 2.- To determine the success rate and incidence of complications in patients with and without side-branch pre-dilation, as well as economic impact in terms of number of used wires.

DETAILED DESCRIPTION:
Introduction: Percutaneous treatment of bifurcation lesion is a complex procedure. After main vessel stent implantation, the side branch became jailed and the carina can be displaced resulting in complete occlusion of this vessel. Re-wiring the side branch in this conditions may result difficult and some times impossible. There is no agreement regarding the need of side branch pre-dilation (before main vessel stent implantation) to reduce these complications. Researchers from European Bifurcation Club have proposed no to pre-dilate the side branch to avoid vessel dissection and difficulties in rewiring the true lumen of the vessel. On the contrary, our group has a good experience in the treatment of bifurcation lesions treated with side branch pre-dilation.

Aims: 1.- To determine the efficacy of the side-branch pre-dilation in patients with bifurcations lesions treated with provisional T stenting. 2.- To determine the success rate and incidence of complications in patients with and without side-branch pre-dilation, as well as economic impact in terms of number of used wires.

Design: Prospective and randomized study. Patients and methods: The series is constituted by 420 patients with bifurcations lesions that will be treated with drug-eluting stents; 210 patients will be treated with side branch pre-dilation before main vessels stent implantation, while the remaining 210 patients will be randomized to no pre-dilation of the side-branch.

Primary end point:

* TIMI flow at Side Branch after main vessel stent implantation.

Secondary end points:

* Time of re-wiring.
* Number of used wires.
* % of stenosis at Side Branch.
* Levels of CK and TpI after the procedure.
* Related cardiac events at 9 months. Relevance: Currently there has been controversy over the use of the side branch pre-dilation in patients with bifurcations lesions treated with provisional T-stenting. However, we have no comparative study in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atherosclerotic coronary disease and bifurcation lesions an significant stenosis of the side branch.
* Main vessels diameter greater than 2.5 mm in diameter at the operator's visual estimate.
* The side branch should exceed 2.25 mm in diameter at the operator's visual estimate.
* Patients with damage to the main branch of any length and the side branch lesions smaller than 5 mm in length.
* Patients with bifurcation lesions fulfilling the following morphologies of the classification of Medina: 1 1 1, 1 0 1, 0 1 1.
* Treatment of bifurcation lesions with previsional drug eluting stents.
* Symptoms of stable angina or acute coronary syndrome.

Exclusion Criteria:

* Contraindication to drug eluting stent implantation.
* Cardiogenic shock.
* Coexistence of other serious systemic diseases.
* Patients in whom it is impossible to guide placement in the side branch before stent implantation in the main vessel.
* Patients with bifurcation lesions and side branch less than 2 mm.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2009-02; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Side branch coronary flow after main vessels stent implantation | Immediately after catheterization procedure

SECONDARY OUTCOMES:
Time required for rewiring of the side branch | Inmediately after catheterization procedure
Number of used wires | Inmediately after catheterization procedure
Levels of markers of myocardial injury (CK and TpI) after the procedure | Immediately after catheterization procedure
Related cardiac events at 9 months | Immediately after catheterization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Pan Alvarez-Osorio, MD, Principal Investigator — Hospital Universitario Reina Sofia de Cordoba
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Córdoba, Spain

REFERENCES:
- [Background] Pan M, Medina A, Suarez de Lezo J, Romero M, Melian F, Pavlovic D, Hernandez E, Segura J, Marrero J, Torres F, et al. Follow-up patency of side branches covered by intracoronary Palmaz-Schatz stent. Am Heart J. 1995 Mar;129(3):436-40. doi: 10.1016/0002-8703(95)90264-3. PMID 7872167
- [Background] Pan M, Suarez de Lezo J, Medina A, Romero M, Hernandez E, Segura J, Castroviejo JR, Pavlovic D, Melian F, Ramirez A, Castillo JC. Simple and complex stent strategies for bifurcated coronary arterial stenosis involving the side branch origin. Am J Cardiol. 1999 May 1;83(9):1320-5. doi: 10.1016/s0002-9149(99)00093-4. PMID 10235088
- [Background] Pan M, Suarez de Lezo J, Medina A, Romero M, Segura J, Ramirez A, Pavlovic D, Hernandez E, Ojeda S, Adamuz C. A stepwise strategy for the stent treatment of bifurcated coronary lesions. Catheter Cardiovasc Interv. 2002 Jan;55(1):50-7. doi: 10.1002/ccd.10057. PMID 11793495
- [Background] Pan M, de Lezo JS, Medina A, Romero M, Segura J, Pavlovic D, Delgado A, Ojeda S, Melian F, Herrador J, Urena I, Burgos L. Rapamycin-eluting stents for the treatment of bifurcated coronary lesions: a randomized comparison of a simple versus complex strategy. Am Heart J. 2004 Nov;148(5):857-64. doi: 10.1016/j.ahj.2004.05.029. PMID 15523318
- [Background] Pan M, Suarez de Lezo J, Medina A, Romero M, Delgado A, Segura J, Ojeda S, Pavlovic D, Ariza J, Fernandez-Duenas J, Herrador J, Urena I. [Six-month intravascular ultrasound follow-up of coronary bifurcation lesions treated with rapamycin-eluting stents: technical considerations]. Rev Esp Cardiol. 2005 Nov;58(11):1278-86. Spanish. PMID 16324581
- [Background] de Lezo JS, Medina A, Pan M, Delgado A, Segura J, Pavlovic D, Melian F, Romero M, Burgos L, Hernandez E, Urena I, Herrador J. Rapamycin-eluting stents for the treatment of unprotected left main coronary disease. Am Heart J. 2004 Sep;148(3):481-5. doi: 10.1016/j.ahj.2004.03.011. PMID 15389236
- [Background] Medina A, Suarez de Lezo J, Pan M. [A new classification of coronary bifurcation lesions]. Rev Esp Cardiol. 2006 Feb;59(2):183. No abstract available. Spanish. PMID 16540043
- [Background] Pan M, Suarez de Lezo J, Medina A, Romero M, Delgado A, Segura J, Ojeda S, Mazuelos F, Hernandez E, Melian F, Pavlovic D, Esteban F, Herrador J. Drug-eluting stents for the treatment of bifurcation lesions: a randomized comparison between paclitaxel and sirolimus stents. Am Heart J. 2007 Jan;153(1):15.e1-7. doi: 10.1016/j.ahj.2006.10.017. PMID 17174630
- [Derived] Pan M, Medina A, Romero M, Ojeda S, Martin P, Suarez de Lezo J, Segura J, Mazuelos F, Novoa J, Suarez de Lezo J. Assessment of side branch predilation before a provisional T-stent strategy for bifurcation lesions. A randomized trial. Am Heart J. 2014 Sep;168(3):374-80. doi: 10.1016/j.ahj.2014.05.014. Epub 2014 Jun 6. PMID 25173550